CLINICAL TRIAL: NCT01709110
Title: Teriparatide and Risedronate in the Treatment of Patients With Severe Postmenopausal Osteoporosis: Comparative Effects on Vertebral Fractures
Brief Title: VERtebral Fracture Treatment Comparisons in Osteoporotic Women
Acronym: VERO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14536; B3D-EW-GHDW (Other: Eli Lilly and Company); 2012-000123-41 (EudraCT Number)
Record Dates: First submitted 2012-10-16; First posted 2012-10-17 (Estimated); Results first posted 2018-01-23 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Postmenopausal Osteoporosis
Keywords: Bone Loss; Vertebral fractures
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Bone Diseases, Metabolic; Spinal Fractures | interventions — Teriparatide; Risedronic Acid; Calcium; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Teriparatide (Experimental): Teriparatide 20 microgram (µg) administered by subcutaneous (SC) injection once daily for 24 months.
  Placebo given orally once weekly for 24 months.
  Elemental Calcium 500 to 1000 milligram per day and Vitamin D 400 to 800 International Units per day, both administered orally once daily while receiving treatment.
  Interventions: Drug: Teriparatide; Drug: Placebo; Drug: Calcium; Drug: Vitamin D
- Risedronate (Active Comparator): Risedronate 35 milligram (mg) administered orally once weekly for 24 months.
  Placebo given by SC injection once daily for 24 months.
  Elemental Calcium 500 to 1000 milligram per day and Vitamin D 400 to 800 International Units per day, both administered orally once daily while receiving treatment.
  Interventions: Drug: Risedronate; Drug: Placebo; Drug: Calcium; Drug: Vitamin D

INTERVENTIONS:
Drug: Teriparatide — Administered SC
  Other Names: LY333334; Forteo; Forsteo
  Arms: Teriparatide
Drug: Risedronate — Administered orally
  Arms: Risedronate
Drug: Placebo — Teriparatide arm placebo administered orally.
  Risedronate arm placebo administered SC.
Drug: Calcium — Administered orally
Drug: Vitamin D — Administered orally

SUMMARY:
The primary purpose of participation in this study is to answer whether teriparatide is superior to risedronate in reducing the occurrence of new vertebral fractures during 24 months of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women with osteoporosis, as defined by low bone mineral density (BMD), i.e. anterior-posterior lumbar spine, total hip or femoral neck BMD ≥1.5 standard deviations below the average BMD for young, healthy, non-Hispanic, Caucasian women
* A minimum of 2 moderate or 1 severe vertebral fragility fractures (confirmed by central reader) were required

Exclusion Criteria:

* Increased risk of osteosarcoma
* History of unresolved skeletal diseases that affect bone metabolism
* History of atypical subtrochanteric or diaphyseal femoral fractures
* Abnormally high or low calcium levels
* Abnormally high parathyroid hormone (PTH) levels
* Severe vitamin D deficiency
* Abnormal thyroid function not corrected by therapy
* History of malignant neoplasms in the last 5 years
* Active liver disease, clinical jaundice
* Significant impairment of hepatic or renal function
* History of nephro- or urolithiasis
* Previous or planned kypho- or vertebroplasty
* Active or risk for osteonecrosis of the jaw
* Active or recent history of upper gastrointestinal disorders
* Unable to stand or sit in the upright position for at least 30 minutes

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1366 (Actual)
Dates: Start 2012-10; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (103):
- United States (30):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Birmingham, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Concord, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fresno, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Laguna Hills, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lancaster, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tustin, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lakewood, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Danbury, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orlando, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gainesville, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Evansville, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Topeka, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bethesda, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Detroit, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Omaha, Nebraska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Clifton, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Freehold, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Albuquerque, New Mexico
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Asheville, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greensboro, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fargo, North Dakota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bend, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Duncansville, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pittsburgh, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wyomissing, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seattle, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Spokane, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madison, Wisconsin
- Argentina (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buenos Aires
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Caba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mar del Plata
- Austria (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Graz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hohenems
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Linz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vienna
- Belgium (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brussels
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Genk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ghent
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gilly
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Laken
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leuven
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Liège
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Merksem
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mons
- Brazil (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brasília
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rio de Janeiro
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., São Paulo
- Canada (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kelowna, British Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vancouver, British Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Halifax, Nova Scotia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamilton, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toronto, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montreal, Quebec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sainte-Foy, Quebec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Trois-Rivières, Quebec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saskatoon, Saskatchewan
- Czechia (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., České Budějovice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Klatovy
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Prague
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Uherské Hradiště
- France (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Caen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Crau
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lyon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orléans
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint-Etienne
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toulouse
- Germany (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dresden
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Frankfurt
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leipzig
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Magdeburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marburg
- Greece (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Athens
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kifissia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pátrai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Thessaloniki
- Hungary (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Budapest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Debrecen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Eger
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kaposvár
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Szeged
- Italy (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Florence
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Genova-Nervi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orbassano
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Padua
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rome
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Torino
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valeggio sul Mincio
- Poland (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bialystok
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Elblag
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lublin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poznan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Świdnik
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan, Puerto Rico
- Spain (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Alzira
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cadiz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sabadell
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valencia

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Body JJ, Marin F, Kendler DL, Zerbini CAF, Lopez-Romero P, Moricke R, Casado E, Fahrleitner-Pammer A, Stepan JJ, Lespessailles E, Minisola S, Geusens P. Efficacy of teriparatide compared with risedronate on FRAX(R)-defined major osteoporotic fractures: results of the VERO clinical trial. Osteoporos Int. 2020 Oct;31(10):1935-1942. doi: 10.1007/s00198-020-05463-4. Epub 2020 May 30. PMID 32474650
- [Derived] Geusens P, Kendler DL, Fahrleitner-Pammer A, Lopez-Romero P, Marin F. Distribution of Prevalent and Incident Vertebral Fractures and Their Association with Bone Mineral Density in Postmenopausal Women in the Teriparatide Versus Risedronate VERO Clinical Trial. Calcif Tissue Int. 2020 Jun;106(6):646-654. doi: 10.1007/s00223-020-00683-6. Epub 2020 Mar 10. PMID 32157334
- [Derived] Minisola S, Marin F, Kendler DL, Geusens P, Zerbini CAF, Russo LA, Casado E, Fahrleitner-Pammer A, Stepan JJ, Lespessailles E, Moericke R, Bagur A, Lakatos P, Lopez-Romero P, Body JJ. Serum 25-hydroxy-vitamin D and the risk of fractures in the teriparatide versus risedronate VERO clinical trial. Arch Osteoporos. 2019 Jan 18;14(1):10. doi: 10.1007/s11657-019-0561-x. PMID 30659410
- [Derived] Geusens P, Marin F, Kendler DL, Russo LA, Zerbini CA, Minisola S, Body JJ, Lespessailles E, Greenspan SL, Bagur A, Stepan JJ, Lakatos P, Casado E, Moericke R, Lopez-Romero P, Fahrleitner-Pammer A. Effects of Teriparatide Compared with Risedronate on the Risk of Fractures in Subgroups of Postmenopausal Women with Severe Osteoporosis: The VERO Trial. J Bone Miner Res. 2018 May;33(5):783-794. doi: 10.1002/jbmr.3384. Epub 2018 Feb 9. PMID 29329484
- [Derived] Kendler DL, Marin F, Zerbini CAF, Russo LA, Greenspan SL, Zikan V, Bagur A, Malouf-Sierra J, Lakatos P, Fahrleitner-Pammer A, Lespessailles E, Minisola S, Body JJ, Geusens P, Moricke R, Lopez-Romero P. Effects of teriparatide and risedronate on new fractures in post-menopausal women with severe osteoporosis (VERO): a multicentre, double-blind, double-dummy, randomised controlled trial. Lancet. 2018 Jan 20;391(10117):230-240. doi: 10.1016/S0140-6736(17)32137-2. Epub 2017 Nov 9. PMID 29129436

RESULTS

PARTICIPANT FLOW:
Groups:
- Teriparatide: Teriparatide 20 microgram (µg) administered by subcutaneous (SC) injection once daily for 24 months.
  Placebo given orally once weekly for 24 months.
- Risedronate: Risedronate 35 milligram (mg) administered orally once weekly for 24 months.
  Placebo given by SC injection once daily for 24 months.
Period: Overall Study
Arm/Group | Teriparatide | Risedronate
Started | 683 | 683
Received at Least One Dose of Study Drug | 680 | 680
Completed | 498 | 515
Not Completed | 185 | 168
Not completed — Adverse Event | 56 | 48
Not completed — Death | 14 | 6
Not completed — Lost to Follow-up | 7 | 5
Not completed — Protocol Violation | 4 | 6
Not completed — Withdrawal by Subject | 96 | 89
Not completed — Physician Decision | 4 | 10
Not completed — Sponsor Decision | 2 | 2
Not completed — Lack of Efficacy | 1 | 1
Not completed — Caregiver Decision | 1 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Teriparatide: Teriparatide 20 microgram administered by subcutaneous injection once daily for 24 months.
  Placebo given orally once weekly for 24 months.
- Risedronate: Risedronate 35 milligram administered orally once weekly for 24 months.
  Placebo given by SC injection once daily for 24 months.
- Total: Total of all reporting groups
Arm/Group | Teriparatide | Risedronate | Total
Number analyzed (Participants) | 680 | 680 | 1360
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.6 (8.77) | 71.6 (8.58) | 72.1 (8.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 680 | 680 | 1360
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 104 | 99 | 203
  Not Hispanic or Latino | 310 | 302 | 612
  Unknown or Not Reported | 266 | 279 | 545
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 4 | 8 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 15 | 20
  White | 670 | 653 | 1323
  More than one race | 0 | 3 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 79 | 78 | 157
  Hungary | 68 | 53 | 121
  Czech Republic | 68 | 68 | 136
  United States | 55 | 67 | 122
  Spain | 66 | 55 | 121
  Greece | 27 | 13 | 40
  Canada | 36 | 33 | 69
  Austria | 24 | 29 | 53
  Belgium | 43 | 45 | 88
  Poland | 55 | 63 | 118
  Brazil | 63 | 81 | 144
  Italy | 33 | 36 | 69
  France | 26 | 29 | 55
  Germany | 37 | 30 | 67
Distribution of Stratification Factors [Count of Participants; unit: Participants] — A participant was considered as having a recent clinical vertebral fragility fracture if she had at least one clinical vertebral fragility fracture within the last 12 months prior to baseline. A participant was considered a recent prior bisphosphonate user if she had received a total of 6 or more months of treatment with any oral bisphosphonate within 3 years prior to baseline.
  Participants
    Vertebral Fracture with Bisphosphonate Use | 82 | 79 | 161
    With Vertebral Fracture without Bisphosphonate Use | 170 | 165 | 335
    Without Vertebral Fracture with Bisphosphonate Use | 184 | 189 | 373
    Without Vertebral Fracture without Bisphosphonate | 244 | 247 | 491
Bone Mineral Density (BMD) [Mean (Standard Deviation); unit: Gram per square centimeter (g/cm2)] — Low BMD is defined as an lumbar spine, total hip or femoral neck BMD ≥ 1.5 standard deviation (SD) below the average BMD for young healthy, non-Hispanic, Caucasian women. Lumbar spine, total hip and femoral neck BMD were assessed by DXA by the investigator at baseline. Population: Any lumbar vertebrae that were not analyzed due to artifacts, fracture, osteophytes, or other abnormalities, should be excluded from the analysis.
  Gram per square centimeter (g/cm2)
    Lumbar Spine: number analyzed (Participants) | 644 | 653 | 1297
    Lumbar Spine | 0.858 (0.1541) | 0.856 (0.1473) | 0.857 (0.1506)
    Femoral Neck: number analyzed (Participants) | 658 | 656 | 1314
    Femoral Neck | 0.662 (0.1085) | 0.667 (0.1129) | 0.664 (0.1107)
    Total Hip: number analyzed (Participants) | 633 | 640 | 1273
    Total Hip | 0.736 (0.1065) | 0.735 (0.1165) | 0.735 (0.1116)
Vertebral Fracture Status [Count of Participants; unit: Participants] — (according to Bioclinica spine x-ray central assessment at baseline).
  Participants
    1 Fracture | 231 | 240 | 471
    2 Fractures | 178 | 174 | 352
    3 Fractures | 104 | 101 | 205
    4 Fractures | 60 | 62 | 122
    5 or More Fractures | 106 | 102 | 208

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With New Vertebral Fractures
Description: The incidence of new vertebral fractures was assessed by quantitative vertebral morphometry measurements (QM) with qualitative visual semiquantitative grading (SQ) confirmation.
  A new vertebral fracture was diagnosed in a vertebra that was non-fractured at the baseline radiological examination. It was defined as a loss of vertebral body height of at least 20% and 4 mm from the baseline radiograph by vertebral QM, based upon placement of six points by a trained, central reader. Any fractures identified by QM were confirmed using SQ: if the vertebral body also had an increase of one or more severity grade, it was considered an incident vertebral fracture.
Time Frame: Baseline through 24 Months
Population: Full analysis set-modified: participants with baseline and at least one post-baseline spinal radiograph evaluable to assess the vertebral fracture status after 24 month of therapy.
Measure: Number; unit: Participants (with at least one event)
Arm/Group | Teriparatide | Risedronate
Number analyzed (Participants) | 516 | 533
Participants (with at least one event) | 28 | 64
Statistical Analysis 1: Comparison: Teriparatide vs Risedronate; Test type: Superiority; p = 0.000094, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test was adjusted for the antecedent of recent clinical vertebral fractures and recent bisphosphonate use; Odds Ratio (OR) = 0.4071, 95% CI 2-sided [0.256 to 0.647]
Statistical Analysis 2: Comparison: Teriparatide vs Risedronate; Test type: Superiority; p = 0.000094, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Risk Ratio (RR) = 0.4431, 95% CI 2-sided [0.290 to 0.677]

2. Secondary Outcome: Proportion of Participants With Pooled New and Worsening Vertebral Fractures
Description: Worsening of a pre-existing fracture was considered if the decrease in vertebral height was at least one severity grade in the semi-quantitative assessment, confirmed by a trained central reader, where vertebrae were graded as normal (SQ0) or as with mild (SQ1), moderate (SQ2), or severe (SQ3) fractures, defined as ~20 to 25% (mild), ~25 to 40% (moderate) or ~40% or more (severe) decrease in anterior, central, or posterior vertebral height (T4 to L4).
Time Frame: Baseline through 24 Months
Population: as for outcome 1
Measure: Number; unit: Participants (with at least one event)
Arm/Group | Teriparatide | Risedronate
Number analyzed (Participants) | 516 | 533
Participants (with at least one event) | 31 | 69
Statistical Analysis 1: Comparison: Teriparatide vs Risedronate; Test type: Superiority; p = 0.000075, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel was adjusted for the antecedent of recent clinical vertebral fractures and recent bisphosphonate use; Odds Ratio (OR) = 0.4187, 95% CI 2-sided [0.269 to 0.652]
Statistical Analysis 2: Comparison: Teriparatide vs Risedronate; Test type: Superiority; p = 0.000075, Cochran-Mantel-Haenszel; [statistical method as in outcome 2, analysis 1]; Risk Ratio (RR) = 0.4561, 95% CI 2-sided [0.305 to 0.682]

3. Secondary Outcome: Proportion of Participants With Pooled Clinical Vertebral and Non-Vertebral Fragility Fractures
Description: A clinical vertebral fracture was defined as a new or worsening vertebral fracture, confirmed by radiography, that was associated with signs and symptoms highly suggestive of a vertebral fracture.
  All non-vertebral fractures that occurred and were diagnosed between visits required the confirmation by the site investigators after evaluating the original x-ray film(s), the radiology or surgical report. For clinical vertebral fractures, the final confirmation of the diagnosis required the centralized evaluation by a trained, independent reader.
Time Frame: Baseline through 24 Months
Population: Full analysis set: all participants who received at least one dose of study drug and had evaluable data.
Measure: Number; unit: Participants (with at least one event)
Arm/Group | Teriparatide | Risedronate
Number analyzed (Participants) | 680 | 680
Participants (with at least one event) | 30 | 61
Statistical Analysis 1: Comparison: Teriparatide vs Risedronate; Test type: Superiority; p = 0.000869, Stratified Log Rank; Stratified Log Rank test was adjusted for the antecedent of recent clinical vertebral fractures and recent bisphosphonate use; Stratified Hazard Ratio (HR) = 0.4831, 95% CI 2-sided [0.316 to 0.739] — The Stratified Hazard Ratio estimate and corresponding 95% CI were obtained from the number of observed and expected events as part of the stratified log-rank test calculations

4. Secondary Outcome: Proportion of Participants With Non-Vertebral Fragility Fractures
Description: A non-vertebral fracture is a fracture at any of the following non-vertebral sites: clavicle, scapula, ribs, sternum, sacrum, coccyx, humerus, radius, ulna, carpus, pelvis, hip, femur, patella, tibia, fibula, ankle, calcaneus, tarsus, and metatarsal. Non-vertebral fractures were determined by direct questioning at each visit, and confirmed by the site investigators by x-ray, radiology or surgical report. Fractures resulting from a severe trauma such as a traffic collision, a beating, or having been struck by a falling or moving object were not considered fragility fractures but traumatic fractures.
Time Frame: Baseline through 24 Months
Population: Full analysis set: all participants who received at least one dose of study drug and had evaluable data.
Measure: Number; unit: Participants (with at least one event)
Arm/Group | Teriparatide | Risedronate
Number analyzed (Participants) | 680 | 680
Participants (with at least one event) | 25 | 38
Statistical Analysis 1: Comparison: Teriparatide vs Risedronate; Test type: Superiority; p = 0.099023, Stratified Log Rank; [statistical method as in outcome 3, analysis 1]; Stratified Hazard Ratio (HR) = 0.6553, 95% CI 2-sided [0.390 to 1.101] — [estimate comment as in outcome 3, analysis 1]

5. Secondary Outcome: Proportion of Participants With Major Non-Vertebral Fragility Fractures
Description: A major non-vertebral fracture is a fracture at any of the following non-vertebral sites hip, radius, humerus, ribs, pelvis, tibia and femur. Non-vertebral fractures were determined by direct questioning at each visit, and confirmed by the site investigators by x-ray, radiology or surgical report. Fractures resulting from a severe trauma such as a traffic collision, a beating, or having been struck by a falling or moving.
Time Frame: Baseline through 24 Months
Population: Full analysis set: all participants who received at least one dose of study drug and had evaluable data.
Measure: Number; unit: Participants (with at least one event)
Arm/Group | Teriparatide | Risedronate
Number analyzed (Participants) | 680 | 680
Participants (with at least one event) | 18 | 31
Statistical Analysis 1: Comparison: Teriparatide vs Risedronate; Test type: Superiority; p = 0.062432, Stratified Log Rank; [statistical method as in outcome 3, analysis 1]; Stratified Hazard Ratio (HR) = 0.5786, 95% CI 2-sided [0.318 to 1.052] — [estimate comment as in outcome 3, analysis 1]

6. Secondary Outcome: Proportion of Participants With New Moderate and/or Severe Vertebral Fractures
Description: Vertebrae were graded as moderate (SQ2), or severe (SQ3) fractures, based on ~25 to 40% (moderate) or ~40% or more (severe) decrease in anterior, central, or posterior vertebral height (T4 through L4).
Time Frame: Baseline through 24 Months
Population: as for outcome 1
Measure: Number; unit: Participants (with at least one event)
Arm/Group | Teriparatide | Risedronate
Number analyzed (Participants) | 516 | 533
Participants (with at least one event) | 26 | 63
Statistical Analysis 1: Comparison: Teriparatide vs Risedronate; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.3812, 95% CI 2-sided [0.237 to 0.614]
Statistical Analysis 2: Comparison: Teriparatide vs Risedronate; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Risk Ratio (RR) = 0.4173, 95% CI 2-sided [0.270 to 0.646]

7. Secondary Outcome: Proportion of Participants With New Multiple (2 or More) Vertebral Fractures
Time Frame: Baseline through 24 Months
Population: as for outcome 1
Measure: Number; unit: Participants (with at least one event)
Arm/Group | Teriparatide | Risedronate
Number analyzed (Participants) | 516 | 533
Participants (with at least one event) | 2 | 12
Statistical Analysis 1: Comparison: Teriparatide vs Risedronate; Test type: Superiority; p = 0.007, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.1593, 95% CI 2-sided [0.035 to 0.728]
Statistical Analysis 2: Comparison: Teriparatide vs Risedronate; Test type: Superiority; p = 0.007, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Risk Ratio (RR) = 0.1643, 95% CI 2-sided [0.036 to 0.744]

8. Secondary Outcome: Proportion of Participants With Pooled Fragility and Traumatic Non-Vertebral Fractures
Description: Traumatic fractures were considered if resulting from a severe trauma such as a traffic collision, a beating, or having been struck by a falling or moving object.
Time Frame: Baseline through 24 Months
Population: Full analysis set: all participants who received at least one dose of study drug and had evaluable data.
Measure: Number; unit: Participants (with at least one event)
Arm/Group | Teriparatide | Risedronate
Number analyzed (Participants) | 680 | 680
Participants (with at least one event) | 40 | 57
Statistical Analysis 1: Comparison: Teriparatide vs Risedronate; Test type: Superiority; p = 0.078, Stratified Log Rank; [statistical method as in outcome 3, analysis 1]; Stratified Hazard Ratio (HR) = 0.6960, 95% CI 2-sided [0.461 to 1.050] — The Stratified Hazard Ratio estimates and corresponding 95% CI were obtained from the number of observed and expected events as part of the stratified log-rank test calculations

9. Secondary Outcome: Change From Baseline to 24 Months Endpoint in Height
Time Frame: Baseline, 24 Months
Population: Full analysis set: all participants who received at least one dose of study drug and had evaluable data.
Measure: Mean (Standard Deviation); unit: Centimeter (cm)
Arm/Group | Teriparatide | Risedronate
Number analyzed (Participants) | 565 | 580
Centimeter (cm)
  Baseline | 154.7 (7.15) | 155.0 (7.40)
  24 Months | 154.3 (7.05) | 154.5 (7.42)
Statistical Analysis 1: Comparison: Teriparatide vs Risedronate; Test type: Superiority; p = 0.093, Mixed Models Analysis — Model included the following fixed effects: treatment, visit, treatment-by-visit interaction, antecedent of recent clinical vertebral fractures, recent use of bisphosphonate and baseline body height(cm); An unstructured covariance matrix was assumed to account for the correlation between observations of the same participant; Least Squares Mean = -0.13, 95% CI 2-sided [-0.28 to 0.02], Standard Error of Mean 0.08 — Treatment difference was calculated as Teriparatide - Risedronate

10. Secondary Outcome: Change From Baseline to 24 Months Endpoint in Back Pain Using an 11-point Numerical Pain Rating Scale
Description: Participants rated the worst back pain during the 24 hours preceding the visit at baseline and each post-baseline visit. An 11-point numerical back pain rating scale (rated from 0 = no back pain to 10 = worst possible back pain) was used.
Time Frame: Baseline, 24 Months
Population: Full analysis set: all participants who received at least one dose of study drug and had evaluable data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Teriparatide | Risedronate
Number analyzed (Participants) | 642 | 648
units on a scale
  Baseline | 4.5 (2.90) | 4.5 (2.91)
  24 Months | 3.4 (2.95) | 3.4 (2.89)
Statistical Analysis 1: Comparison: Teriparatide vs Risedronate; Test type: Superiority; p = 0.585, Mixed Models Analysis — Model included the following fixed effects: treatment, visit, treatment-by-visit interaction, antecedent of recent clinical vertebral fractures, recent use of bisphosphonate and baseline back pain (no pain - worst pain [0-10]); [statistical method as in outcome 9, analysis 1]; Least Squares Mean = -0.09, 95% CI 2-sided [-0.42 to 0.24], Standard Error of Mean 0.17 — Treatment difference was calculated as Teriparatide - Risedronate

11. Secondary Outcome: Change From Baseline to 24 Months Endpoint in the European Quality of Life Questionnaire [EQ-5D-5L] (UK)
Description: The EQ-5D-5L is a generic, multidimensional, health-related, quality-of-life instrument completed on five dimensions to measure health-related quality of life. The profile allowed participants to rate their health state in five health domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression using a five level scale (no problems, slight problems, moderate problems, severe problems, and unable to/extreme problems). The responses are used to derive the health state index scores using the United Kingdom (UK) algorithm, with scores ranging from -0.59 to 1.0. A higher score indicates better health state.
Time Frame: Baseline, 24 Months
Population: Full analysis set: all participants who received at least one dose of study drug and had evaluable data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Teriparatide | Risedronate
Number analyzed (Participants) | 642 | 647
units on a scale
  Baseline | 0.59 (0.243) | 0.62 (0.228)
  24 Months | 0.65 (0.249) | 0.68 (0.205)
Statistical Analysis 1: Comparison: Teriparatide vs Risedronate; Test type: Superiority; p = 0.757, Mixed Models Analysis — Model included the following fixed effects: treatment, visit, treatment-by-visit interaction, antecedent of recent clinical vertebral fractures, recent use of bisphosphonate baseline EQ-5D-5L (UK); [statistical method as in outcome 9, analysis 1]; Least Squares Mean = -0.00, 95% CI 2-sided [-0.03 to 0.02], Standard Error of Mean 0.01 — Treatment difference was calculated as Teriparatide - Risedronate

12. Secondary Outcome: Change From Baseline to 24 Months Endpoint in the European Quality of Life Questionnaire [EQ-5D-5L] (US)
Description: The EQ-5D-5L is a generic, multidimensional, health-related, quality-of-life instrument completed on five dimensions to measure health-related quality of life. The profile allowed participants to rate their health state in five health domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression using a five level scale (no problems, slight problems, moderate problems, severe problems, and unable to/extreme problems). The responses are used to derive the health state index scores using the United States (US) cross walk algorithm, with scores ranging from -0.11 to 1.0. A higher score indicates better health state.
Time Frame: Baseline, 24 Months
Population: Full analysis set: all participants who received at least one dose of study drug and had evaluable data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Teriparatide | Risedronate
Number analyzed (Participants) | 642 | 647
units on a scale
  Baseline | 0.70 (0.167) | 0.72 (0.159)
  24 Months | 0.74 (0.176) | 0.76 (0.145)
Statistical Analysis 1: Comparison: Teriparatide vs Risedronate; Test type: Superiority; p = 0.694, Mixed Models Analysis — Model included the following fixed effects: treatment, visit, treatment-by-visit interaction, antecedent of recent clinical vertebral fractures, recent use of bisphosphonate baseline EQ-5D-5L (US); [statistical method as in outcome 9, analysis 1]; Least Squares Mean = -0.00, 95% CI 2-sided [-0.02 to 0.01], Standard Error of Mean 0.01 — Treatment difference was calculated as Teriparatide - Risedronate

ADVERSE EVENTS:
Arm/Group | Teriparatide | Risedronate
Serious Adverse Events (participants affected / at risk) | 138/683 | 117/683
Other Adverse Events (participants affected / at risk) | 130/683 | 130/683
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Teriparatide (N=683) | Risedronate (N=683)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pernicious anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 3 (3) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 5 (5) | 3 (3)
Atrioventricular block (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 2 (2) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac valve disease (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tricuspid valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricle outflow tract obstruction (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Goitre (Endocrine disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Femoral hernia, obstructive (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal achalasia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatic cyst (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 1 (1)
Regurgitation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (2) | 0 (0)
Performance status decreased (General disorders) | 1 (1) | 0 (0)
Sudden cardiac death (General disorders) | 0 (0) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 2 (2)
Ischaemic hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Abdominal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 3 (3) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Escherichia pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (2) | 3 (3)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 3 (3)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Pyonephrosis (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (3) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Craniocerebral injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 15 (16) | 19 (21)
Femoral neck fracture (Injury, poisoning and procedural complications) | 4 (4) | 3 (3)
Femur fracture (Injury, poisoning and procedural complications) | 3 (4) | 6 (7)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 5 (5)
Humerus fracture (Injury, poisoning and procedural complications) | 3 (3) | 5 (5)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 3 (4) | 6 (6)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Post procedural stroke (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural vomiting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Rib fracture (Injury, poisoning and procedural complications) | 3 (4) | 1 (3)
Scapula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 2 (6) | 3 (4)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Blood pressure increased (Investigations) | 1 (1) | 0 (0)
Carbohydrate antigen 19-9 increased (Investigations) | 0 (0) | 1 (1)
General physical condition abnormal (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (5)
Kyphosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Periostitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chondrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cystadenocarcinoma ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hypergammaglobulinaemia benign monoclonal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebellar ischaemia (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral artery embolism (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Embolic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1)
Intercostal neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 2 (2) | 3 (3)
Multiple sclerosis (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Radicular pain (Nervous system disorders) | 1 (1) | 1 (1)
Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 2 (2) | 0 (0)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 3 (3) | 2 (2)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 2 (2)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Vascular dementia (Nervous system disorders) | 1 (1) | 0 (0)
Vascular encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Device dislocation (Product Issues) | 1 (1) | 0 (0)
Device malfunction (Product Issues) | 0 (0) | 1 (1)
Alcohol abuse (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 1 (1)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 2 (2)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Female genital tract fistula (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Uterine prolapse (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Systemic lupus erythematosus rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0)
Arterial disorder (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 3 (3)
Granulomatosis with polyangiitis (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 2 (2)
Hypertensive crisis (Vascular disorders) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 4 (4) | 0 (0)
Peripheral artery occlusion (Vascular disorders) | 1 (1) | 0 (0)
Subclavian artery occlusion (Vascular disorders) | 0 (0) | 1 (1)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Teriparatide (N=683) | Risedronate (N=683)
Arthralgia (Musculoskeletal and connective tissue disorders) | 44 (54) | 51 (63)
Back pain (Musculoskeletal and connective tissue disorders) | 73 (77) | 79 (89)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 37 (45) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days